CLINICAL TRIAL: NCT02444507
Title: A Randomized, Two-Way Crossover, Single-Dose Pharmacokinetic Study to Evaluate the Bioequivalence of a Test Formulation Compared to an Equivalent Dose of a Reference Drug Product (Nexium Powder for Injection and Infusion 40 mg) in Healthy Adult Subjects
Brief Title: A Pharmacokinetic Study to Evaluate the Bioequivalence of a Test Formulation Compared to an Equivalent Dose of a Reference Drug Product
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: isRed Pharma & Biotech Research Corporation (Industry)
Collaborators: Yung Shin Pharmaceutical Ind. Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: YSP RFH3002-01
Record Dates: First submitted 2015-05-08; First posted 2015-05-14 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Injections; Solutions

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Reference Drug: Nexium (Active Comparator): Name: Nexium powder for injection and infusion 40 mg, Active substance: Esomeprazole 40 mg, Each single dose of esomeprazole 40 mg will be administrated as intravenous infusion over 30 minutes.
  Interventions: Drug: Nexium powder for injection and infusion 40 mg
- Test Drug: Esomelone (Active Comparator): Name: Esomelone Powder for Solution for Injection / Infusion 40 mg Active substance: Esomeprazole 40 mg, Each single dose of esomeprazole 40 mg will be administrated as intravenous infusion over 30 minutes.
  Interventions: Drug: Esomelone Powder for Solution for Injection / Infusion 40 mg

INTERVENTIONS:
Drug: Nexium powder for injection and infusion 40 mg — Reference Drug, Active substance: Esomeprazole 40 mg, Each single dose of esomeprazole 40 mg will be administrated as intravenous infusion over 30 minutes.
  Arms: Reference Drug: Nexium
Drug: Esomelone Powder for Solution for Injection / Infusion 40 mg — Test Drug, Active substance: Esomeprazole 40 mg, Each single dose of esomeprazole 40 mg will be administrated as intravenous infusion over 30 minutes.
  Arms: Test Drug: Esomelone

SUMMARY:
To assess the bioequivalence of esomeprazole of the TEST product vs. the REFERENCE product in healthy volunteers who reside in Taiwan.

DETAILED DESCRIPTION:
This study is designed to assess the bioequivalence of esomeprazole of the TEST product vs. the REFERENCE product in healthy volunteers who reside in Taiwan. Bioequivalence will be assumed if the 90% confidence interval of the AUC0-t, AUC0-inf and Cmax ratio are within the 80-125% interval for log-transformed values.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, aged between 20 to 40 years old.
2. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests, chest x-ray and electrocardiogram.
3. The normal range of the body mass index should between 18.5 and 25.
4. Normal laboratory determinations results including: SGOT (AST), SGPT (ALT), albumin, glucose, creatinine, uric acid, cholesterol, TG, γ-GT, alkaline phosphatase, total bilirubin, BUN, HBsAg, Anti-HCV and Anti-HIV test.
5. Normal hematology results including: hemoglobin, hematocrit, WBC count with differential, RBC count and platelet count.
6. Normal urinalysis results including: glucose, protein, RBC, WBC, epith, casts and bacteria.
7. Female subject who is:

   * using adequate contraception since last menstruation and no plan for conception during the study.
   * non-lactating.
   * has negative pregnancy test (urine) within 14 days prior to the study.
8. Informed consent form signed.

Exclusion Criteria:

1. A history of drug or alcohol abuse during the past 24 weeks.
2. Sensitivity to analogous drug.
3. A clinically significant illness (such as significant unintentional weight loss, recurrent vomiting, dysphagia, haematemesis, melaena or gastric ulcer) within the past 4 weeks.
4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoetic, neurological, pulmonary or gastrointestinal pathology within the past 4 weeks.
5. Planed vaccination during the time course of the study.
6. Participation of any clinical investigation during the last 60 days.
7. Regular use of any medication during the last 4 weeks.
8. Single use of any medication during the last 2 weeks.
9. Blood donation of more than 250 mL within the past 12 weeks.
10. Individuals are judged by the investigator or co-investigator to be undesirable as subjects.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-05 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence will be assumed if the 90% confidence interval of the AUC0-t, AUC0-inf and Cmax ratio are within the 80-125% interval for log-transformed values. | Sampling Schedule: 0, 0.167, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10 and 12 hr
  The calculation of the respective pharmacokinetic will be based upon the reported concentrations and sampling times.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan